CLINICAL TRIAL: NCT05824676
Title: Utility of the Variable Angle LCP Patella Plating System for Traumatic Patellar Fractures: A Randomized Control Trial
Brief Title: DePuy Synthes Variable Angle LCP Patella Plating System Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Michael Miranda, Clinical Professor, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHC-2022-0283
Record Dates: First submitted 2023-03-01; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-02

CONDITIONS: Trauma; Patella Fracture; Knee Cap; Knee Cap Injury; Knee Discomfort; Knee Deformity
Keywords: Patella; Plating; trauma; kneecap; injury; knee injuries; knee injury; fracture; break; randomized
MeSH Terms: conditions — Wounds and Injuries; Patella Fracture; Knee Injuries; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant
Masking Description: It insures unbiased patient reported outcomes in data collection, the participants are blinded to what arm they are put in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Depuy Synthes LCP Patella Plating System (Experimental): This group will have 18 randomly selected participants, who will receive the Depuy Synthes LCP Patella Plating System for patella fracture.
  Interventions: Device: Variable Angle LCP Patella Plating System
- Control/Conventional Fixation (Other): This group will have 18 randomly selected participants, who will receive the conventional treatment for patella fracture.
  Interventions: Device: Traditional Fixation

INTERVENTIONS:
Device: Variable Angle LCP Patella Plating System — FDA approved device, 510K number of, K210408. The Variable Angle LCP Patella Plating System is a device that can be formed to a patients specific need with various anchoring points to best fix what is needed for fixation.
  Arms: Depuy Synthes LCP Patella Plating System
Device: Traditional Fixation — Traditional fixation methods for patellar fracture (screws, suture fixation, wire fixation, other plates).
  Arms: Control/Conventional Fixation

SUMMARY:
The Depuy Synthes Locking Compression Plate (LCP) Variable Angle Patella Plating System is an FDA approved device. The purpose of this study is to see how well the Depuy Synthes LCP Variable Plating System work in fixing a broken kneecap (patella). Depuy says that the device will improve healing when compared to traditional ways of repairing a broken patella.

The goal of this randomized control trial is to learn how well the LCP Variable Plating System works to fix a broken patella (kneecap) compared to traditional fixation methods, in male and females, age 18 to 74, with a patellar fracture, and being treated at Hartford HealthCare The Bone and Joint Institute or Hartford Hospital. The main question it aims to answer are:

* To understand if the Depuy Synthes LCP Variable Angle Plating System will provide a better way to help patients recover from a broken patella.

Participants will evaluated at specific time points: post-op day 1, 6 weeks, 3 months, 6 months, and 12 month post-surgery. Participants will be asked to:

* Complete surveys at all evaluation timepoints.
* Have x-rays(radiographs) taken at the 6 week, 3 month, 6 month, 9 month, and 1 year timepoints.
* Participants will have a passive range of motion tests done at 6 week, 3 month, 6 month, 9 month, and 1 year timepoints.
* Participants would have strength and balance tests done at the 3 month, 6 month, 9 month, and 1 year timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age between 18 and 74 years old (inclusive)
* Patellar fracture
* Treated at Hartford HealthCare The Bone and Joint Institute or Hartford Hospital

Exclusion Criteria:

* Age greater than or equal to 75 or less than 18
* Patients that are non-ambulatory/limited ambulation prior to their injury
* Previous patellar fracture
* Pre-existing osteoarthritis of the knee
* Ipsilateral femoral or tibia fractures

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
DePuy Synthes LCP Variable Angle Patella Plating System clinical outcomes comparison | 1 year
  Comparing the DePuy Synthes LCP Variable Patella Plating System to tradition fixation methods using clinical outcomes measures.
DePuy Synthes LCP Variable Angle Patella Plating System functional outcomes comparison | 1 year
  Comparing the DePuy Synthes LCP Variable Patella Plating System to traditional fixation methods using functional outcomes measures.
DePuy Synthes LCP Variable Angle Patella Plating System patient reported outcomes comparison | 1 year
  Comparing the DePuy Synthes LCP Variable Angle Patella Plating System to traditional fixation methods using patient/participant reported outcomes measures.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System 10 Global (PROMIS 10 Global) | Post-op day 1
  PROMIS Global-10 is a validated 10-question survey used to assess health care-related quality of life measures such as a participant's function, mental health, numeric pain scale for the general population. The scale runs from 0 to 20. 0 represents severe impairment and low quality of life. A score of 20 represents the best possible quality of life.
Patient-Reported Outcomes Measurement Information System 10 Global (PROMIS 10 Global) | 6 weeks
  PROMIS Global-10 is a validated 10-question survey used to assess health care-related quality of life measures such as a participant's function, mental health, numeric pain scale for the general population. The scale runs from 0 to 20. 0 represents severe impairment and low quality of life. A score of 20 represents the best possible quality of life.
Patient-Reported Outcomes Measurement Information System 10 Global (PROMIS 10 Global) | 3 months
  PROMIS Global-10 is a validated 10-question survey used to assess health care-related quality of life measures such as a participant's function, mental health, numeric pain scale for the general population. The scale runs from 0 to 20. 0 represents severe impairment and low quality of life. A score of 20 represents the best possible quality of life.
Patient-Reported Outcomes Measurement Information System 10 Global (PROMIS 10 Global) | 6 months
  PROMIS Global-10 is a validated 10-question survey used to assess health care-related quality of life measures such as a participant's function, mental health, numeric pain scale for the general population. The scale runs from 0 to 20. 0 represents severe impairment and low quality of life. A score of 20 represents the best possible quality of life.
Patient-Reported Outcomes Measurement Information System 10 Global (PROMIS 10 Global) | 9 months
  PROMIS Global-10 is a validated 10-question survey used to assess health care-related quality of life measures such as a participant's function, mental health, numeric pain scale for the general population. The scale runs from 0 to 20. 0 represents severe impairment and low quality of life. A score of 20 represents the best possible quality of life.
Patient-Reported Outcomes Measurement Information System 10 Global (PROMIS 10 Global) | 1 year
  PROMIS Global-10 is a validated 10-question survey used to assess health care-related quality of life measures such as a participant's function, mental health, numeric pain scale for the general population. The scale runs from 0 to 20. 0 represents severe impairment and low quality of life. A score of 20 represents the best possible quality of life.
Activities of Daily Living-Knee Outcomes Survey (ADL-KOS) | Post-op day 1
  ADL-KOS is a 14 question survey that assesses a participant's functional ability related to their knee and how knee symptoms may affect their activities of daily living. The scoring for the ADL-KOS runs from 0 to 100. 0 representing the lowest possible functional ability, and 100 representing the maximum functional ability possible.
Activities of Daily Living-Knee Outcomes Survey (ADL-KOS) | 6 weeks
  ADL-KOS is a 14 question survey that assesses a participant's functional ability related to their knee and how knee symptoms may affect their activities of daily living. The scoring for the ADL-KOS runs from 0 to 100. 0 representing the lowest possible functional ability, and 100 representing the maximum functional ability possible.
Activities of Daily Living-Knee Outcomes Survey (ADL-KOS) | 3 months
  ADL-KOS is a 14 question survey that assesses a participant's functional ability related to their knee and how knee symptoms may affect their activities of daily living. The scoring for the ADL-KOS runs from 0 to 100. 0 representing the lowest possible functional ability, and 100 representing the maximum functional ability possible.
Activities of Daily Living-Knee Outcomes Survey (ADL-KOS) | 6 months
  ADL-KOS is a 14 question survey that assesses a participant's functional ability related to their knee and how knee symptoms may affect their activities of daily living. The scoring for the ADL-KOS runs from 0 to 100. 0 representing the lowest possible functional ability, and 100 representing the maximum functional ability possible.
Activities of Daily Living-Knee Outcomes Survey (ADL-KOS) | 9 months
  ADL-KOS is a 14 question survey that assesses a participant's functional ability related to their knee and how knee symptoms may affect their activities of daily living. The scoring for the ADL-KOS runs from 0 to 100. 0 representing the lowest possible functional ability, and 100 representing the maximum functional ability possible.
Activities of Daily Living-Knee Outcomes Survey (ADL-KOS) | 1 year
  ADL-KOS is a 14 question survey that assesses a participant's functional ability related to their knee and how knee symptoms may affect their activities of daily living. The scoring for the ADL-KOS runs from 0 to 100. 0 representing the lowest possible functional ability, and 100 representing the maximum functional ability possible.
Radiographs | 6 weeks
  Radiographic imaging will be taken at each of the study visits starting at week 6 to assess healing and ensure that there are no issues with the hardware. Radiographic healing will be assessed by the congruity of the cortical bone and reduction of fracture lines. Radiographs will also be used to determine if there is any failure of the hardware. (i.e. loosening of the screws or wires or instrument breakage).
Radiographs | 3 months
  Radiographic imaging will be taken at each of the study visits starting at week 6 to assess healing and ensure that there are no issues with the hardware. Radiographic healing will be assessed by the congruity of the cortical bone and reduction of fracture lines. Radiographs will also be used to determine if there is any failure of the hardware. (i.e. loosening of the screws or wires or instrument breakage).
Radiographs | 6 months
  Radiographic imaging will be taken at each of the study visits starting at week 6 to assess healing and ensure that there are no issues with the hardware. Radiographic healing will be assessed by the congruity of the cortical bone and reduction of fracture lines. Radiographs will also be used to determine if there is any failure of the hardware. (i.e. loosening of the screws or wires or instrument breakage).
Radiographs | 9 months
  Radiographic imaging will be taken at each of the study visits starting at week 6 to assess healing and ensure that there are no issues with the hardware. Radiographic healing will be assessed by the congruity of the cortical bone and reduction of fracture lines. Radiographs will also be used to determine if there is any failure of the hardware. (i.e. loosening of the screws or wires or instrument breakage).
Radiographs | 1 year
  Radiographic imaging will be taken at each of the study visits starting at week 6 to assess healing and ensure that there are no issues with the hardware. Radiographic healing will be assessed by the congruity of the cortical bone and reduction of fracture lines. Radiographs will also be used to determine if there is any failure of the hardware. (i.e. loosening of the screws or wires or instrument breakage).
Passive Range of Motion (ROM) | 6 weeks
  Passive ROM will be assessed at each study visit starting at 6 weeks. Knee flexion and extension will be measured using a goniometer (an instrument that measures angles of joints). Participants will be asked to sit with their hips at 90° and lower leg hanging off the exam table or chair. The center of the goniometer will be placed at the rotational axis of the knee joint and the two arms of the goniometer will be aligned with the femoral shaft and tibial shaft. The participant's leg will then be maximally flexed and the goniometer read to determine the total flexion range, and then the participant's leg will be straightened to determine the maximum extension angle. The total knee arc of motion will be recorded as the addition of these two angles.
Passive Range of Motion (ROM) | 3 months
  Passive ROM will be assessed at each study visit starting at 6 weeks. Knee flexion and extension will be measured using a goniometer (an instrument that measures angles of joints). Participants will be asked to sit with their hips at 90° and lower leg hanging off the exam table or chair. The center of the goniometer will be placed at the rotational axis of the knee joint and the two arms of the goniometer will be aligned with the femoral shaft and tibial shaft. The participant's leg will then be maximally flexed and the goniometer read to determine the total flexion range, and then the participant's leg will be straightened to determine the maximum extension angle. The total knee arc of motion will be recorded as the addition of these two angles.
Passive Range of Motion (ROM) | 6 months
  Passive ROM will be assessed at each study visit starting at 6 weeks. Knee flexion and extension will be measured using a goniometer (an instrument that measures angles of joints). Participants will be asked to sit with their hips at 90° and lower leg hanging off the exam table or chair. The center of the goniometer will be placed at the rotational axis of the knee joint and the two arms of the goniometer will be aligned with the femoral shaft and tibial shaft. The participant's leg will then be maximally flexed and the goniometer read to determine the total flexion range, and then the participant's leg will be straightened to determine the maximum extension angle. The total knee arc of motion will be recorded as the addition of these two angles.
Passive Range of Motion (ROM) | 9 months
  Passive ROM will be assessed at each study visit starting at 6 weeks. Knee flexion and extension will be measured using a goniometer (an instrument that measures angles of joints). Participants will be asked to sit with their hips at 90° and lower leg hanging off the exam table or chair. The center of the goniometer will be placed at the rotational axis of the knee joint and the two arms of the goniometer will be aligned with the femoral shaft and tibial shaft. The participant's leg will then be maximally flexed and the goniometer read to determine the total flexion range, and then the participant's leg will be straightened to determine the maximum extension angle. The total knee arc of motion will be recorded as the addition of these two angles.
Passive Range of Motion (ROM) | 1 year
  Passive ROM will be assessed at each study visit starting at 6 weeks. Knee flexion and extension will be measured using a goniometer (an instrument that measures angles of joints). Participants will be asked to sit with their hips at 90° and lower leg hanging off the exam table or chair. The center of the goniometer will be placed at the rotational axis of the knee joint and the two arms of the goniometer will be aligned with the femoral shaft and tibial shaft. The participant's leg will then be maximally flexed and the goniometer read to determine the total flexion range, and then the participant's leg will be straightened to determine the maximum extension angle. The total knee arc of motion will be recorded as the addition of these two angles.
Strength | 3 months
  Quadriceps muscle strength will be assessed starting at each visit starting at the 3 month post-operative visit. Strength measures will be assessed using a hand held dynamometer (a device that measures force). The strength assessment will be performed with the participant in a seated position with hips at 90°. The dynamometer will be placed mid tibial shaft and the testers other hand will be placed just above the knee to provide stability. The participant will be instructed to try to straighten their leg against the resistance of the examiner. The strength measures will be repeated 3 times for consistency. Additionally, the strength of the non-injured quadriceps will also be assessed to determine if there is a side to side strength deficit.
Strength | 6 months
  Quadriceps muscle strength will be assessed starting at each visit starting at the 3 month post-operative visit. Strength measures will be assessed using a hand held dynamometer (a device that measures force). The strength assessment will be performed with the participant in a seated position with hips at 90°. The dynamometer will be placed mid tibial shaft and the testers other hand will be placed just above the knee to provide stability. The participant will be instructed to try to straighten their leg against the resistance of the examiner. The strength measures will be repeated 3 times for consistency. Additionally, the strength of the non-injured quadriceps will also be assessed to determine if there is a side to side strength deficit.
Strength | 9 months
  Quadriceps muscle strength will be assessed starting at each visit starting at the 3 month post-operative visit. Strength measures will be assessed using a hand held dynamometer (a device that measures force). The strength assessment will be performed with the participant in a seated position with hips at 90°. The dynamometer will be placed mid tibial shaft and the testers other hand will be placed just above the knee to provide stability. The participant will be instructed to try to straighten their leg against the resistance of the examiner. The strength measures will be repeated 3 times for consistency. Additionally, the strength of the non-injured quadriceps will also be assessed to determine if there is a side to side strength deficit.
Strength | 1 year
  Quadriceps muscle strength will be assessed starting at each visit starting at the 3 month post-operative visit. Strength measures will be assessed using a hand held dynamometer (a device that measures force). The strength assessment will be performed with the participant in a seated position with hips at 90°. The dynamometer will be placed mid tibial shaft and the testers other hand will be placed just above the knee to provide stability. The participant will be instructed to try to straighten their leg against the resistance of the examiner. The strength measures will be repeated 3 times for consistency. Additionally, the strength of the non-injured quadriceps will also be assessed to determine if there is a side to side strength deficit.
Balance | 3 months
  Balance assessments will also take place at each visit starting at the 3 month post-operative visit. Static balance will be assessed using a portable force plate. Participants will be asked to perform four balance tasks. The first will be with both feet together hands on their hips staring straight ahead. The second assessment will be both feet together, hands on their hips with their eyes closed. The final two assessments will be single limb stances with eyes open. One single limb stance will be used to assess the operative limb the other the non-operative limb. Each balance task will be measured for 20 seconds. During this time investigator will record the medial lateral weight shift, anterior posterior weight shift, and sway area, a 90% elliptical fit of the weight shift with the minor and major axes defined as the maximum and minimum sway values in anterior/posterior and medial/lateral directions.
Balance | 6 months
  Balance assessments will also take place at each visit starting at the 3 month post-operative visit. Static balance will be assessed using a portable force plate. Participants will be asked to perform four balance tasks. The first will be with both feet together hands on their hips staring straight ahead. The second assessment will be both feet together, hands on their hips with their eyes closed. The final two assessments will be single limb stances with eyes open. One single limb stance will be used to assess the operative limb the other the non-operative limb. Each balance task will be measured for 20 seconds. During this time investigator will record the medial lateral weight shift, anterior posterior weight shift, and sway area, a 90% elliptical fit of the weight shift with the minor and major axes defined as the maximum and minimum sway values in anterior/posterior and medial/lateral directions.
Balance | 9 months
  Balance assessments will also take place at each visit starting at the 3 month post-operative visit. Static balance will be assessed using a portable force plate. Participants will be asked to perform four balance tasks. The first will be with both feet together hands on their hips staring straight ahead. The second assessment will be both feet together, hands on their hips with their eyes closed. The final two assessments will be single limb stances with eyes open. One single limb stance will be used to assess the operative limb the other the non-operative limb. Each balance task will be measured for 20 seconds. During this time investigator will record the medial lateral weight shift, anterior posterior weight shift, and sway area, a 90% elliptical fit of the weight shift with the minor and major axes defined as the maximum and minimum sway values in anterior/posterior and medial/lateral directions.
Balance | 1 year
  Balance assessments will also take place at each visit starting at the 3 month post-operative visit. Static balance will be assessed using a portable force plate. Participants will be asked to perform four balance tasks. The first will be with both feet together hands on their hips staring straight ahead. The second assessment will be both feet together, hands on their hips with their eyes closed. The final two assessments will be single limb stances with eyes open. One single limb stance will be used to assess the operative limb the other the non-operative limb. Each balance task will be measured for 20 seconds. During this time investigator will record the medial lateral weight shift, anterior posterior weight shift, and sway area, a 90% elliptical fit of the weight shift with the minor and major axes defined as the maximum and minimum sway values in anterior/posterior and medial/lateral directions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford HealthCare The Bone and Joint Institute, Hartford, Connecticut, United States